CLINICAL TRIAL: NCT05921643
Title: Short- and Medium-term Evaluation of Mastoid Filling Using Bioactive Glass"
Acronym: GLASS-BONA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: GLASS-BONA
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cholesteatoma
MeSH Terms: conditions — Cholesteatoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with cholesteatoma who has never been operated on: All patients will benefit from surgical management for a first stage cholesteatoma in the operating room under general anesthesia. The surgical technique (closed technique) is the reference technique for the management of cholesteatoma in adults. It involves a cartilaginous removal to reconstruct the attical region. Then a filling material is used to fill the mastoid (GlassBONE™ or Bonalive™), and above all to stabilize the cartilaginous fragment to prevent a recurrence. The mastoid filler used is left to the discretion and habits of the surgeon.
  Interventions: Device: verre bioactif 45S5 GlassBONE; Device: verre bioactif S53P4 Bonalive

INTERVENTIONS:
Device: verre bioactif 45S5 GlassBONE — All patients will benefit from surgical management for a first stage cholesteatoma in the operating room under general anesthesia. The surgical technique (closed technique) is the reference technique for the management of cholesteatoma in adults. It involves a cartilaginous removal to reconstruct the attical region. Then a filling material is used to fill the mastoid (GlassBONE™ or Bonalive™), and above all to stabilize the cartilaginous fragment to prevent a recurrence. The mastoid filler used is left to the discretion and habits of the surgeon.
Device: verre bioactif S53P4 Bonalive — All patients will benefit from surgical management for a first stage cholesteatoma in the operating room under general anesthesia. The surgical technique (closed technique) is the reference technique for the management of cholesteatoma in adults. It involves a cartilaginous removal to reconstruct the attical region. Then a filling material is used to fill the mastoid (GlassBONE™ or Bonalive™), and above all to stabilize the cartilaginous fragment to prevent a recurrence. The mastoid filler used is left to the discretion and habits of the surgeon.

SUMMARY:
Adult patients referred to the ENT surgery department of the Hospices Civils de Lyon with cholesteatoma that had never been operated on.

All patients will benefit from surgical management for cholesteatoma initially in the operating room under general anesthesia. The surgical technique (closed technique) is the reference technique for the management of cholesteatoma in adults. It involves a cartilaginous removal to reconstruct the attical region. Then a filling material is used to fill the mastoid (GlassBONE™ or Bonalive™), and above all to stabilize the cartilaginous fragment to prevent a recurrence.

DETAILED DESCRIPTION:
Patients are operated on as an outpatient and receive a phone call the next morning to look for an initial complication. The patients will be reviewed in consultation at D8, D45, 3 months, 6 months and at 18 months with clinical examination (otoscopy) and audiometry at each consultation. The consultation on D8 is used for removal of the expandable cotton put in place in the external auditory canal (CAE) during surgery to guide healing, control post-auricular healing and look for signs of complication during the examination. A cone beam (CBCT) is performed during the consultation on D45 to confirm the correct position of the ossiculoplasty and check the persistence of the initial filling. The proportion of filled mastoid at D45 will serve as a reference to then be compared to the CT scan at 6 months and at 18 months. During surgery, and at the consultation at 6 months and 18 months, patients will also have to complete a quality of life questionnaire (Chronic Ear Survey French version; in the Appendix).

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old
* Patients with proven cholesteatoma
* Patient requiring and agreeing to surgery with filling of the mastoid or tympanic epi (closed technique with filling)
* Patient having a surgery with filling in first intention

Exclusion Criteria:

* Background:
* Known outer, middle or inner ear malformation
* Congenital cholesteatoma
* Previously operated cholesteatoma
* Cholesteatoma requiring an open technique or presenting with chronic non-cholesteatomatous otitis
* Contraindications to the use of GlassBONE™ or Bonalive™
* Pregnant, parturient or nursing mothers
* Persons deprived of their liberty by a judicial or administrative decision, persons subject to psychiatric care, adults subject to a measure of legal protection or unable to express themselves
* Patient participating in interventional research excluding routine care research (old regulations) and category 2 research that does not interfere with the analysis of the primary endpoint
* Patient objecting to the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients referred to the ENT surgery department of the Hospices Civils de Lyon with cholesteatoma that had never been operated on.
  All patients will benefit from surgical management for cholesteatoma initially in the operating room under general anesthesia. The surgical technique (closed technique) is the reference technique for the management of cholesteatoma in adults. It involves a cartilaginous removal to reconstruct the attical region. Then a filling material is used to fill the mastoid (GlassBONE™ or Bonalive™), and above all to stabilize the cartilaginous fragment to prevent a recurrence.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
mastoid filling | 6 month
  A patient will be considered as a responder if the proportion of mastoid filling at 6 months is strictly greater than 70% compared to the reference measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud, Lyon, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No